CLINICAL TRIAL: NCT06360718
Title: Effects of a Storybook About New Leukemia Diagnosis Versus Standard Child Life Intervention on Parental Stress: a Pilot Randomized Controlled Study
Brief Title: Effects of Using a Storybook, to Explain Leukemia to Children Versus the Standard Child Life Intervention, on Parental Stress.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Erin Shields, Child Life Specialist III, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHLA-23-00170
Record Dates: First submitted 2024-04-03; First posted 2024-04-11 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Leukemia
Keywords: Parental stress; Diagnosis education; Leukemia; Child life; Cancer; Chemotherapy; Hair Loss; School-Age; Intervention; Family-Centered Care
MeSH Terms: conditions — Leukemia; Neoplasms; Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Parents in this group will receive the standard child life interventional support for explaining the leukemia diagnosis to the school-aged patient/sibling. Parents in this study will complete surveys at three timepoints, these surveys include: (1) Comfort Survey (prior to child life intervention), (2) Discharge Survey (about 1 week following the child life intervention), and the (3) Parenting Stress Index-4-Short Form (at baseline, at the time of the discharge survey, and about 3.5 months later).
- Intervention (Storybook) Group (Experimental): Parents in this group will receive the "Who is Luke Eemia?" storybook, and will receive guidance from the child life specialist on how to utilize the storybook with their school-aged child. Parents in this study will complete surveys at three timepoints, these surveys include: (1) Comfort Survey (prior to child life intervention), (2) Discharge Survey and (3) Storybook Assessment survey to review the parent's impression of the storybook intervention tool (about 1 week following the child life intervention), and the (4) Parenting Stress Index -4-Short Form (at baseline, at the time of the discharge survey, and about 3.5 months later).
  Interventions: Behavioral: "Who is Luke Eemia?" Storybook

INTERVENTIONS:
Behavioral: "Who is Luke Eemia?" Storybook — Parents in this group will receive the "Who is Luke Eemia?" storybook, and will receive guidance from the child life specialist on how to utilize the storybook with their school-aged child. Parents in this study will complete surveys at three timepoints, these surveys include: (1) Comfort Survey (prior to child life intervention), (2) Discharge Survey and (3) Storybook Assessment survey to review the parent's impression of the storybook intervention tool (at the time of discharge, or about 1 week following the child life intervention), and the (4) Parenting Stress Index -4-Short Form (at baseline, at the time of the discharge survey, and about 3.5 months later).
  Arms: Intervention (Storybook) Group

SUMMARY:
The goal of this clinical trial is to measure the effects of using a storybook versus standard child life intervention with parents of children newly diagnosed with leukemia on parental stress.

The main questions it aims to answer are:

* What effect will the storybook have on parent/legal guardian stress at three timepoints: baseline, discharge, and follow up?
* Will this storybook impact parent/legal guardian comfort levels and improve their child's understanding?

Participants will be asked to complete surveys at three timepoints, prior to and following child life intervention and about 3.5 months later. During child life interventions, participants will receive resources and support to explain leukemia to their school aged, 3-16-year-old, child (patient or sibling).

Researchers will compare Intervention and Control Groups to see if parental stress is lower in those who received the storybook in addition to the standard child life intervention versus the standard child life intervention alone.

DETAILED DESCRIPTION:
Research Design:

This is a pilot randomized controlled study.

Control Group will receive the standard child life care and interventions following a new leukemia diagnosis. This includes meeting one of the primary hematology oncology inpatient certified child life specialists (CCLS) to discuss patient/sibling understanding, language used, family experiences or stressors, and family goals when disclosure information about the diagnosis. Interventions may include books about cancer, personalized learning stories, or interactive activities to explain leukemia, cancer, and chemotherapy.

Intervention Group will receive the standard child life care described in the Control Group above, plus the "Who Is Luke Eemia?" Storybook intervention tool created for this study. This storybook was designed by the PI to offer education on leukemia, cancer, chemotherapy, and hair loss through a child life lens. The CCLS will introduce the storybook and discuss common developmental considerations, offering parents suggestions on how to use it with their child, and answer additional questions.

Study Procedures:

70 Parent/Child Dyads will be enrolled in this study.

The study team will screen patients upon admission to the inpatient unit, identifying patients newly diagnosed with leukemia. Eligibility criteria requires a patient or sibling to be English or Spanish speaking, and between the ages of 3-16 years of age (without any cognitive or developmental delays or chronic medical conditions). Parent participation requires child assent to enroll.

Enrolled parents will be randomized in the storybook group (intervention), or the standard child life support (control). The school-aged children will be enrolled as research subjects, though all study measures will be completed by parents, including parental impression of their child's understanding.

To assess the effects of the storybook intervention tool, versus the standard child life intervention, parents will complete surveys at three timepoints:

Baseline:

* Parenting Stress Index Short Form (PSI™-4-SF)
* Comfort Survey

Discharge:

* Discharge Survey
* Storybook Assessment (Intervention Group Only)
* The Parenting Stress Index Short Form (PSI™-4-SF)

Follow Up (about 3.5 months after Baseline):

- The Parenting Stress Index Short Form (PSI™-4-SF)

Summary statistics means, medians, standard deviations and interquartile range will be calculated to summarize variables, we will trend data using graphs, and we will perform pre planned statistical tests in R.

ELIGIBILITY:
Parents are approached and enrolled on the inpatient Hematology Oncology unit at CHLA, during the admission where their child received a new leukemia diagnosis.

Inclusion Criteria:

* Parent/Legal Guardian of a child a. who is school-aged (3-16 years old) with a new leukemia diagnosis b. with a new leukemia diagnosis who is not school-aged but is a sibling of a school-aged child (<3 years or >16 years old).
* Parent/legal guardian is able to speak, read, and write English or Spanish, and give informed consent 3. Parent/legal guardian is over 18 years of age.

Exclusion Criteria:

* Their school-aged children have developmental or cognitive delays, and/or other chronic illnesses.
* Their school-aged child does not give assent to participate.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-02-03 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Parental Stress, prior to and following child life intervention | 10 minutes at each timepoint (30 minutes total over the study).
  All participating parents/legal guardians will be given the Parenting Stress Index -4 Short Form [PSI™-4-SF] at baseline (before child life intervention), discharge (about 1 week following the child life intervention for extended admissions), and about 3.5 months after the initial survey. The PSI™-4-SF form is a 36-item scale, available in English and Spanish. The form is broken into two domains (child and parent). The questions in the Parent Domain look at identifying sources of stress.

SECONDARY OUTCOMES:
Parent's Comfort Explaining Aspects of Leukemia Diagnosis | at Baseline
  All parents/legal guardians will be given the Comfort Survey to assess parent comfort levels and parent perception of their child's understanding of the leukemia diagnosis prior to receiving the child life intervention. The Comfort Survey is a non-standardized survey, designed by the PI to elicit information about parental comfort explaining the diagnosis at baseline
Parental Impression of the Storybook Tool using a Likert scale (1-week post baseline). | Baseline to 1 week
  Parents/legal guardians randomized to the Intervention Group will complete the Storybook Assessment survey. The Storybook Assessment will measure the parent's overall impression of the educational storybook intervention tool.
Parent perception of the child's stress | 10 minutes at each timepoint (30 minutes total over the study).
  All participating parents/legal guardians will be given the PSI™-4-SF at baseline (before child life intervention), discharge (about 1 week following the child life intervention for extended admissions), and about 3.5 months after the initial survey. The PSI™-4-SF form is a 36-item scale, available in English and Spanish. The form is broken into two domains (child and parent). The Child Domain will explore questions around the parent's perception of the child's stress.
Parent comfort, readiness, and importance, explaining aspects of the diagnosis at the discharge (1-week post baseline). | Baseline to 1 week
  All parents/legal guardians will be given the Discharge Survey to assess the parent's perceived importance, comfort, and readiness around discussing aspects of the diagnosis with their child at the time of discharge (about 1 week following the child life intervention). The Discharge Survey will elicit information about their comfort and readiness to explain the diagnosis following child life intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Shields, MA, Principal Investigator — Children's Hospital Los Angeles; Kaitlin Bennett, Principal Investigator — Children's Hospital Los Angeles; Mandy Flores, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No